CLINICAL TRIAL: NCT05705206
Title: Feasibility and Accuracy of Core Temperature Measurements Using the Esophageal Temperature Probe Inserted Through the Gastric Lumen of Supraglottic Airway Device in Pediatrics: a Prospective Observational Study
Brief Title: Feasibility and Accuracy of Core Temperature Measurements Using the Esophageal Temperature Probe Inserted Through the Gastric Lumen of Supraglottic Airway Device in Pediatrics
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hajung Kim, Clinical assistant professor, Asan Medical Center
Other Study IDs: 2020-1695
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Temperature Change, Body; Supraglottic Airway Device; Pediatric ALL
MeSH Terms: conditions — Body Temperature Changes; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In pediatric patients, the accuracy of body temperature measured with an esophageal temperature probe placed through the gastric lumen of the supraglottic airway device is investigated.

DETAILED DESCRIPTION:
Pediatric patients using a supraglottic airway device during general anesthesia are targeted. When the patient enters the operating room, standard monitoring is performed, general anesthesia is induced, a supraglottic airway device is installed, and an anesthesiologist inserts an esophageal thermometer through the gastric lumen. We recorded the body temperature measured in the esophagus, tympanic membrane, temporal artery, and rectum every 10 minutes from 10 minutes after insertion.

ELIGIBILITY:
Inclusion Criteria:

* Pediatrics patients under six years old with ASA PS 1-3
* Patients undergoing general anesthesia using the Supraglottic airway device
* Patient's weight: 10-30kg

Exclusion Criteria:

* Patients who refused to participate in the study
* Patients with tumors in the esophagus or esophageal varices
* Patients with a monitoring device inserted through the esophagus during surgery
* Patients with ear inflammation
* Patients with congenital anomaly in the rectum
* Patients judged unfit to participate in the study by medical staff for other reasons

Max Age: 6 Years | Sex: All
Age Groups: Child
Study Population: Pediatrics patients under six years old patients undergoing general anesthesia using the Supraglottic airway device
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Comparison of esophageal temperature and temperature at tympanic membrane, rectum, temporal artery | 10min
  'c

SECONDARY OUTCOMES:
Effect of gastric suction through an esophageal temperature probe | After inserting the esophageal temperature probe
  Evaluated via gastric sonography

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided